CLINICAL TRIAL: NCT05688787
Title: Efficacy of Perineural Injection Therapy in a Group of Egyptians Patients With Primary Fibromyalgia: Non-Randomized Controlled Study
Brief Title: Efficacy of Perineural Injection Therapy in Primary Fibromyalgia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mervat Eissa, Associate Professor, Cairo University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PerineuralFMS
Record Dates: First submitted 2023-01-09; First posted 2023-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Fibromyalgia, Primary
Keywords: Perineural Injection
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Intervention Model Description: The participants in intervention group will be received 4 sessions of perineural injection
  1 week a part with optional additional sessions per the physician recommadation and the patient preference. other group, will be received standard of care treatment of fibromyalgia
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Perineural injection arm (Active Comparator): 30 patients will be received 4 sessions of perineural injection
  1 week a part with optional additional sessions per the physician recommadation and the patient preference .injections are done with a 27 gauge half 1/2 needle directed perpendicular to the skin and going
  1/ to the skin surface delivering 1_2 cc of buffered 5% dextrose solution in the subcutaneous superficial perineural tissue we will be targeting the most triggering points for each patient emphasizing on pain located in thoraco-dorsal fascia, the fascia of the erectorspinae muscles along T10 to L2 dorsal rami, interspinoustenderness from medial branches of dorsal rami, superiorcluneal nerve at 7-8 cm from middle line cross the iliac crest & T10 cross over iliac crest at a distance 8-10cm
  Interventions: Procedure: Perineural Injection
- Standard treatment (No Intervention): will be received standard of care treatment of fibromyalgia

INTERVENTIONS:
Procedure: Perineural Injection — .injections are done with a 27 gauge half 1/2 needle directed perpendicular to the skin and going
  1/ to the skin surface delivering 1_2 cc of buffered 5% dextrose solution in the subcutaneous superficial perineural tissue we will be targeting the most triggering points for each patient emphasizing on pain located in thoraco-dorsal fascia, the fascia of the erectorspinae muscles along T10 to L2 dorsal rami, interspinoustenderness from medial branches of dorsal rami, superiorcluneal nerve at 7-8 cm from middle line cross the iliac crest& T10 cross over iliac crest at a distance 8-10cm
  Arms: Perineural injection arm

SUMMARY:
The goal of fibromyalgia Treatment is to relieve the pain and improve quality of life and physical function which need a

Final Version: April 2019Research Template 3 multifaceted treatment approach involving non pharmacological pain management and medicine

Lyftgot perineural injection therapy "lyftgot PIT" previously known as neural prolotherapy , is a method of injection treatment designed and developed by DR Lyftgot from new Zealand to treat the neurogenic inflammation and the neuropathic pain caused by the sensocrine small nerve fiber .PIT is based on the injection of small amount of dextrose 5%in a neutral PH sterile water solution in the subcutaneous tissue around the sick nerve to correct the neuroglycopenia and to inhibit the neurogenic inflammation.

DETAILED DESCRIPTION:
Fibromyalgia is a chronic non inflammatory wide spread pain disorder associated with a complex of symptoms as fatigue, depression and cognitive impairment , it is the second most common disorder encountered in rheumatology practice (Berger et aL,2007) The pathophysiology is certainly unclear involves a number of factors , including abnormalities in the neuroendocrine and autonomic nervous system ,psychological variables, genetic factor, and environmental stressors (Hudson JI, 2006 ) Fibromyalgia is no longer a diagnosis of exculsion ,patient are diagnosed according to the American college of rheumatology diagnostic criteria which requires a three conditions to be met a wide spread pain index >7 and symptom severity scale score >5 or WPI from 3-6 and ss scale score >9, symptoms have been present at similar level for at least 3 month and patient doesn't have a disorderthat would otherwise explain the pain

The goal of fibromyalgia Treatment is to relieve the pain and improve quality of life and physical function which need a

Final Version: April 2019Research Template 3 multifaceted treatment approach involving non pharmacological pain management and medicine

Lyftgot perineural injection therapy "lyftgot PIT" previously known as neural prolotherapy , is a method of injection treatment designed and developed by DR Lyftgot from new Zealand to treat the neurogenic inflammation and the neuropathic pain caused by the sensocrine small nerve fiber .PIT is based on the injection of small amount of dextrose 5%in a neutral PH sterile water solution in the subcutaneous tissue around the sick nerve to correct the neuroglycopenia and to inhibit the neurogenic inflammation These small nerve fibers are responsible for delivering to the tissue the nerve growth factors necessary for the repair healing and reconstruction of the connective tissue system connecting the superficial skin system to the deep myo-fascial-skeletal system and for restoration of its original compostion with its normal osmotic and electro magnetic pressure (lyftogt,2007) Dextrose 5% block the TRPV1 receptor which inhibit the propagation of the neuropathic pain signal giving the patient the immediate analgesia , it also inhibit the neurogenic inflammation and stimulate the release of nerve growth factor that help in thr repair PIT is a novel , safe, effective and economical treatment for the pain felt in fibromyalgia In this study we aim to asses the efficacy of this treatment in alleviating the pains felt by these patients

ELIGIBILITY:
Inclusion Criteria:.

* Adult fully conscious patients fulling the American college of rheumatology preliminary diagnostic criteria for fibromyalgia

Exclusion Criteria:

* Any other causes of secondary fibromyalgia or musculoskeletal pain as osteoarthritis , endocrinal disease (thyroid dysfunction)
* Rheumatic MSK diseases commonly associated with secondary fibromyalgia as rheumatoid arthritis, SLE
* less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Fibromyalgia impact questionnaire | 3 moths
  assessment of the quality of life and function
visual analogue scale | 3 months
  visual analogue scale, numeric rating scale for measuring the pain

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alainy Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided